CLINICAL TRIAL: NCT02583113
Title: A Retrospective Consecutive Series Patient Preference and Clinical Outcomes Study in Bilateral Knee Osteoarthritis Patients With Both Total Knee Arthroplasty and Unicompartment Knee Arthroplasty Prostheses.
Brief Title: Bilateral Total Knee Arthroplasty vs Unicompartment Arthroplasty Retrospective and Clinical Outcome Study
Status: Withdrawn | Type: Observational
Why Stopped: Alternate Research Pursued
Sponsor: Medacta USA (Industry)
Responsible Party: Sponsor
Other Study IDs: UNI 001
Record Dates: First submitted 2015-10-20; First posted 2015-10-21 (Estimated); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Osteoarthritis
Keywords: Total Knee Replacement; Unicompartment Knee Replacement
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Total and Unicompartment Knee Replacement
  Interventions: Device: Total and Unicompartment Knee Replacement

INTERVENTIONS:
Device: Total and Unicompartment Knee Replacement — Patients who have undergone a primary TKA on one side and primary UKA on the opposite side and are at a minimum of two years post-surgery.
  Other Names: TKA UKA

SUMMARY:
To determine if there is a patient satisfaction preference of Total Knee Arthroplasty (TKA) vs Unicompartmental Knee Arthroplasty (UKA) in patients with bilateral knee osteoarthritis who underwent a primary TKA one side and a primary UKA on the opposite side and are at a minimum of two years post-surgery. Patient reported outcomes and data with be analyzed along with all retrospective chart data.

ELIGIBILITY:
Inclusion Criteria:

1. Must be able to read, understand and provide written informed consent on the Institutional Review Board (IRB) approved Informed Consent Form (ICF)
2. Ability to understand and provide written authorization for use and disclosure of personal health information
3. Subject who are able and willing to comply with the study protocol and follow-up visit
4. Must be 18 years or older to participate
5. Subjects must have a clinically documented osteoarthritis in both knees, single or multiple compartments
6. Subjects must have undergone a primary TKA and primary UKA in the contralateral knee
7. Must be a minimum 2 year (24 months) post-surgery on each knee
8. One or both TKA/UKA surgeries must have been performed by the Principal Investigator.
9. Subjects must be able to return for the follow-up appointment, and have the mental capacity to cooperate with PRO's, questionnaires, physical exam and radiographs

Exclusion Criteria:

1. Subjects who underwent UKA with Patella Femoral Joint (PFJ) replacement on the same side.
2. Women who are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients that have undergone a Total Knee and Unicompartment knee replacement contralateral.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-02; Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate patient preference of Total Knee Arthroplasty (TKA) vs Unicompartmental Knee Arthroplasty (UKA) | Minimum 2 years post surgery
  Asking patients "which is your better knee overall"

SECONDARY OUTCOMES:
Knee Injury and Osteoarthritis Outcome Score (KOOS) | Minimum 2 years post-op
  Knee symptoms, pain, function, and QoL
Forgotten Joint Score (FJS) | Minimum of 2 years post-op
  Knee function-patient's ability to forget the artificial joint in everyday life
Knee Society Score (KSS) subjective measures | Minimum of 2 years post-op
  Patient Expectation and Satisfaction Sub-scores
Euro-Qual Health Related Quality of Life (EQ-5D) | Minimum of 2 years post-op
  General health status
Return to work history | Minimum of 2 years post-op
  Questionnaire for work history prior to surgery and after surgery
Radiographic Analysis | Pre-operative and minimum of 2 years post-op
  Radiographic analysis will include evaluation of component and limb alignment, evidence of component subsidence or migration, and the presence and progression of radiolucent lines between the prosthesis, bone and cement.
Knee Society Score (KSS) Objective measures | Minimum of 2 years post-op
Demographics | Pre-operative and Minimum of 2 years post-op

OTHER OUTCOMES:
Complications will be recorded | Pre-operative and minimum 2 years post-operative

CONTACTS AND LOCATIONS:
Overall Officials: Mukesh Ahuja, MBBS, MS, Study Director — Medacta USA, Inc
Locations (1):
- Tri County Orthopeadic Center, Leesburg, Florida, United States